CLINICAL TRIAL: NCT03162211
Title: Improving Outcomes of Depression Through Person-centered Measurement-based Care and Individualized Feedback
Brief Title: Feedback to Improve Depression Outcomes
Acronym: PCMBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1022385; Catalyst 1160 (Other Grant/Funding Number: Nova Scotia Health Research Foundation)
Record Dates: First submitted 2017-04-25; First posted 2017-05-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback Arm (Experimental): A registry platform including access to all self-report rating scales and the feedback mechanism will be made available to all patients. Patients in the experimental group will receive automated reminders (by text message, phone and/or email) to complete outcome measures each week. Feedback forms will be comprehensive and condensed to a one page report including graphical presentations of symptom course and text. Clinician feedback forms will include content on depression severity over time and recommendations for individualized treatment. Patient feedback forms will also incorporate depression severity over time as well as summary information on achievement towards personalized treatment goals. The intervention will last 6-months, with feedback forms being generated once per week for the first three month and then each month for a total of fifteen feedback time points. Patients in the feedback group will be encouraged to meet with their clinician each month to discuss the feedback.
  Interventions: Other: Feedback Report
- No Feedback Arm (No Intervention): A registry platform including access to all self-report rating scales and the feedback mechanism will be made available to all patients. Patients in the control group will not receive regular reminders or be sent feedback reports on an automatic regular basis.

INTERVENTIONS:
Other: Feedback Report — There are two types of feedback forms: 1. Patient feedback forms and 2. Clinician feedback forms. Feedback form content has been developed in consultation with a board of clinicians, service providers, and patients living with depression. Feedback forms will be comprehensive and condensed to a one page report including graphical presentations of symptom course and text. Clinician feedback forms will include content on depression severity over time and recommendations for individualized treatment. Patient feedback forms will also incorporate depression severity over time as well as summary information on achievement towards personalized treatment goals.
  Arms: Feedback Arm

SUMMARY:
Depression is a leading cause of burden in Canada and globally. Although more people now seek and receive treatment for depression, there are still many who do not respond well to treatments. New and low-cost options are needed to improve the lives of people with depression. Research suggests that asking patients to complete questionnaires and sending feedback to their clinicians may improve depressive symptoms. Research also shows that encouraging individuals with depression to take part in shaping their own care can be beneficial. To date, no research has examined a combination of these two approaches. This project aims to investigate the benefits of providing personalized feedback to patients and clinicians in order to improve the care and outcomes for people with depression in Canada. To answer this research question, adults who are diagnosed with depression will be placed in one of two groups: 1. The patient and clinician will receive feedback to help guide further care based on the patient's responses to questionnaires 2. The patient and clinician will not receive feedback. The feedback form has been developed with input from clinicians, researchers and people with lived experience of depression, and follows new Canadian treatment guidelines. Information including depressive symptoms, quality of life, personal goals for recovery, and healthcare costs will be collected for a year or longer using an online data collection platform. The research team includes clinician-scientists, healthcare managers, educators, primary care physician and people with lived experience of depression. This project has the potential to deliver significant health benefits for individuals with depression, lessen the population burden of depression and improve the health care system by optimizing care delivery and improving quality of life at low cost.

DETAILED DESCRIPTION:
Goal: To improve the outcomes of depression by applying measurement based care that is person-centered and provides individualised feedback to providers and patients within a collaborative mental health care framework.

Background: Depression is a leading cause of disease burden in Canada and globally. Although help-seeking and treatment rates have increased, the outcomes of depression remain unsatisfactory with high rates of inadequate treatment response, chronicity and recurrence. Recent data suggest that measurement-based care with regular ratings of depression symptoms coupled with feedback of results to clinicians and patients may improve outcomes. There is also evidence for the benefits of person-centered approaches that empower individuals living with depression to take active part in shaping their care. Person-centered care that integrates measurement-based feedback is yet to be tested.

Aims: To test the benefits of person-centered measurement-based care in improving outcomes of depression in contemporary Canadian primary and collaborative health care context.

Approach: We will test the benefits of person-centered measurement-based feedback in a randomized registry trial. Adults aged 18 or older diagnosed with major depressive disorder or persistent depressive disorder will be allocated to have a regular measurement-based feedback sent to themselves and their clinicians or not in a 1:1 ratio. The feedback was designed with a council of individuals with depression following the principles of patient-centered and measurement-based care and the recommendations of the 2016 Canadian Network for Mood and Anxiety Treatment guidelines. An on-line registry platform will be used to collect self-report and clinician-rated depression severity, role functioning, quality of life and person-centered self-defined goals. The primary outcome will be meaningful change in treatment and depression severity measured with the self-reported Quick Inventory of Depressive Symptomatology at 1, 3, 6 and 12 months after study entry. Secondary measures will include remission of depression, core role and occupational functioning, quality of life, healthcare cost and self-defined treatment goals. A cost-effectiveness analysis will determine the cost of improved outcomes in terms of quality of life.

Core expertise: The applicants include clinician-scientists, healthcare managers, educators and people with lived experience of depression. The applicants have expertise in depression, primary and collaborative care, clinical trials, epidemiology, statistics, psychometrics and health economics. The registry and feedback forms were developed as part of the Canadian Depression Research and Intervention Network which promotes involvement of individuals with lived experience in research. The database and statistical analyses are supported by the Research Methods Unit.

Expected outcomes: This project will deliver an innovative platform for person-centered measurement-based care for depression through collaborative mental health care. We expect that person-centered measurement-based care will lead to significant health benefits by optimizing care delivery, reducing burden of depression and improving quality of life at low cost. The outcomes of this research will be disseminated through professional networks, patient support organizations, on-line media and education of health professionals.

ELIGIBILITY:
Inclusion criteria:

* a diagnosis of MDD or PDD established with the Structured Clinical Interview for DSM-5 (SCID-5)
* depression being the primary current problem requiring clinical attention judged by an intake clinician
* age 18 or more (no upper limit)
* capacity to provide informed consent

Exclusion criteria:

* lifetime diagnosis of bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective disorder, current alcohol or drug use disorder
* pregnancy
* acute suicide risk (Montgomery and Asberg Depression Rating Scales (MADRS) (suicide item≥4)
* current psychotic symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Meaningful change in treatment | Month 0-6
  The first primary outcome will be a meaningful change in treatment as assessed by a clinical expert using CANMAT guidelines.
Total score QIDS-SR | Month 0-6
  The second primary outcome will be the total score ranging from 0-27 on the 16-item QIDS-SR, a widely used and extensively validated self-report measure of depressive symptoms that aligns closely with DSM diagnostic criteria for depression.

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | Month 0-6
  Secondary outcomes include the MADRS completed by a clinical researcher blind to allocation
WSAS | Month 0-6
  Core role and occupational functioning as measured by the total score on the self-report 5-item Work and the Social Adjustment Scales (WSAS)
LEAPS | Month 0-6
  Core role and occupational functioning as measured by the total score on the self-report 11-item Lam Employment Absence and Productivity Scale (LEAPS).
EQ-5D | Month 0-6
  Health-related quality of life will be measured with the EQ-5D.32 The EQ-5D measures the extent to which an individual's health impacts quality of life and is recommended for Canadian economic evaluations.
My Top Goal | Month 0-6
  Self-defined treatment goals will be measured by My Top Goal, personalized in content (individual's most valued treatment goal) and standardized in scale (0-100% goal achievement).

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Uher, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No